CLINICAL TRIAL: NCT04042506
Title: In Situ Vaccination With Stereotactic Body Radiation Therapy (SBRT) as a Strategy to Overcome Resistance to Immune Checkpoint Blockade: a Phase II Clinical Trial of SBRT and Anti-PD-1 Therapy With Immunologic Correlates
Brief Title: SBRT as a Vaccination for Metastatic Melanoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Unable to enroll patients in this study
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J18145; IRB00188445 (Other: JHM IRB)
Record Dates: First submitted 2019-07-31; First posted 2019-08-02 (Actual); Last update posted 2021-04-12 (Actual); Status verified 2020-04

CONDITIONS: Metastatic Melanoma
Keywords: immune checkpoint blockade; SBRT; Nivolumab
MeSH Terms: conditions — Melanoma | interventions — Nivolumab; Radiosurgery

STUDY DESIGN:
Intervention Model Description: This is a single-institution, single-arm phase II study. SBRT will be given to a single extracranial metastatic site in combination with nivolumab.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Extracranial SBRT and Nivolumab (Experimental): Stereotactic body radiation therapy (SBRT) will be given to a single extracranial metastatic site in combination with nivolumab.
  Patients will receive nivolumab 480mg intravenously (IV) every 4 weeks (1 cycle = 8 weeks), as well as SBRT dose of 8-10 Gy x 3 fractions (at maximum 3 doses per week) delivered to 1 extracranial site between days 1-14 of Cycle 1.
  Nivolumab will be continued until confirmed progression, unacceptable toxicity, or total of 6 Cycles (whichever occurs first).
  Interventions: Drug: Nivolumab 10 MG/ML Intravenous Solution [OPDIVO]; Radiation: Stereotactic Body Radiation Therapy (SBRT)

INTERVENTIONS:
Drug: Nivolumab 10 MG/ML Intravenous Solution [OPDIVO] — 480mg IV every 4 weeks
  Other Names: Opdivo
Radiation: Stereotactic Body Radiation Therapy (SBRT) — SBRT dose of 8-10 Gy x 3 fractions (at maximum 3 doses per week) delivered to 1 extracranial site between days 1-14 of Cycle 1.

SUMMARY:
Immunotherapy with PD-1 blockade is a first-line treatment for patients with advanced melanoma, but unfortunately most patients progress on this therapy. Recent evidence suggests that radiation can enhance the immune response in the presence of checkpoint blockade. The investigators aim to determine if radiation can elicit increased immune responses in patients who have stable or progressive disease on nivolumab.

DETAILED DESCRIPTION:
To determine safety of stereotactic body radiation therapy (SBRT) in presence of ICB in patients with advanced unresectable melanoma. Toxicity will be deemed acceptable if the rate of Grade 3+ adverse events (CTC v4) is ≤ 33%, with relevant AEs defined as either of the following occurring between the start of SBRT and 12 weeks following SBRT completion:

* Any grade 3-5 metabolic or hematological toxicity that is related, probably related or possibly related to nivolumab or SBRT.
* Any grade 3-5 non-hematological toxicity that is related, probably related or possibly related to SBRT.

Secondary Endpoints:

• To determine whether SBRT results in a clinical abscopal effect on unirradiated lesions. The hypothesized rate of abscopal effect is >14%.

Exploratory Correlative studies:

* In select patients for whom TCRseq reveals clonal expansion in non-irradiated tumor and serial blood specimens, the relevance of such expansion to tumor-specific responses will be investigated using mutation-associated neoantigens (MANAFEST) assays.
* Serial stool specimens will be studied to correlate potential changes in microbiome with abscopal effect.
* To determine whether SBRT promotes clonal expansion of melanoma-specific T-cells, in both peripheral blood and within TME of non-irradiated lesions.
* To determine whether TCR clonal expansion correlates with clinically observed abscopal response.
* To identify additional immunological biomarkers in the non-irradiated (abscopal) TME using intratumoral gene expression profiling to assess for induction and upregulation of a Type I IFN signature among responders1-3. IHC in TME will be used to characterize modulation of immune cell populations pre- and post-SBRT, and to assess correlation of PD-L1 and other immune-checkpoint receptor expression with responsiveness to SBRT and changes in TME post-SBRT.

ELIGIBILITY:
Inclusion Criteria:

* Signed Written Informed Consent
* Willing and able to provide informed consent
* Age ≥ 18 years
* Target Population
* Histological confirmation of melanoma
* Advanced unresectable (AJCC Stage III or IV) disease (cutaneous, mucosal, acral or ocular)
* Stable disease or progression (RECIST 1.1) after anti-PD-1 monotherapy (≥ 16 weeks and ≥ 2 CT assessments). The maximum time period off anti-PD-1 monotherapy, prior to protocol therapy, cannot exceed 2 months.
* Prior systemic treatment regimen in the advanced/metastatic setting is allowed (BRAF inhibitor, chemotherapy, cytokine/biologic therapy or clinical trial)
* Prior treatment with anti-CTLA-4 checkpoint inhibitor is allowed
* Minimum of 2 or more measurable lesions by RECIST 1.1, with at least 1 lesion accessible for clinical, US, or CT-guided needle biopsy. If 2 lesions, then one of those must measure 4cm in maximum diameter and be amenable for biopsy; this lesion will be utilized for abscopal effect determination as well. Otherwise, if 3 or more lesions are present, one lesion will receive SBRT, 2nd lesion will be used for radiographic abscopal response assessment, and 3rd lesion will be used for pre- and post-treatment biopsies.
* ECOG Performance Status of 0-1

Exclusion Criteria:

* Target Disease Exceptions
* Prior radiation within 6 months of enrollment (excluding brain metastases), or at any time to one of the 3 lesions for treatment/assessment
* If patient has >1 lesion which requires immediate/urgent management with RT due to present or impending clinical consequences (uncontrolled pain, risk of loss of function), such a patient will not be enrolled on this trial
* Medical History and Concurrent Diseases

  * Major toxicity from prior anti-PD-1 which precludes continuation of anti-PD-1 therapy.
  * Pregnancy or inability to use contraception (if childbearing age)
  * Any active or recent history of a known or suspected autoimmune disease or recent history of a syndrome that required systemic corticosteroids (> 10 mg daily prednisone equivalent) or immunosuppressive medications except for syndromes which would not be expected to recur in the absence of an external trigger. Subjects with vitiligo or type I diabetes mellitus or residual hypothyroidism due to autoimmune thyroiditis only requiring hormone replacement are permitted to enroll. Patients with psoriasis not requiring active, systemic treatment are allowed.
  * Any condition requiring systemic treatment with corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days prior to first dose of study drug. Inhaled steroids and adrenal replacement steroid doses up to 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease
  * Uncontrolled adrenal insufficiency
  * Requirement for anti-coagulation with Coumadin, low molecular weight heparin and anti-thrombin inhibitors will be accepted if anticoagulation has been stable for at least 4 weeks and no recent history of prior bleeding complications.
  * Prior malignancy active within the previous 3 years except for locally curable cancers that have been apparently cured such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the cervix, breast or low risk Gleason 6 prostate cancer
  * Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS); Any positive test for hepatitis B or hepatitis C virus indicating acute or chronic infection
  * Known medical condition (e.g., a condition associated with diarrhea or acute diverticulitis) that, in the investigator's opinion, would increase the risk associated with study participation or study drug administration or interfere with the interpretation of safety results
  * Major surgery (i.e., nephrectomy) less than 28 days prior to the first dose of study drug
  * Anti-cancer therapy less than 14 days prior to the first dose of study drug or palliative, focal radiation therapy less than 14 days prior to the first dose of study drug
  * Presence of any toxicities attributed to prior immunotherapy, other than alopecia, that have not resolved to Grade 1 (NCI CTCAE v4) or baseline before administration of study drug
* Physical and Laboratory Test Findings: Any of the following laboratory test findings:

  * WBC < 2,000/mm3
  * Neutrophils < 1,500/mm3
  * Platelets < 100,000/mm3
  * AST or ALT > 3 x ULN (> 5 x ULN if liver metastases are present)
  * Total Bilirubin > 1.5 x ULN (except subjects with Gilbert Syndrome, who can have total bilirubin < 3.0 mg/dL)
  * Serum creatinine > 1.5 x upper limit of normal (ULN) or creatinine clearance < 40 mL/min (measured or calculated by Cockroft-Gault formula)
* Allergies and Adverse Drug Reaction: History of severe hypersensitivity reaction to any monoclonal antibody or study drug components
* Other Exclusion Criteria

  * Prisoners or subject who are involuntarily incarcerated
  * Not suitable for SBRT treatment
  * Subjects who are compulsorily detained for treatment of either a psychiatric or physical illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-11-26 (Actual); Primary Completion 2019-11-26 (Actual); Study Completion 2021-01-26 (Actual)

PRIMARY OUTCOMES:
Safety of SBRT in the presence of immune checkpoint blockade (ICB) as measured by number of participants experiencing adverse events | 12 weeks
  Number of participants with advanced unresectable melanoma, receiving SBRT in the presence of ICB who experience metabolic or hematological, or non-hematological adverse events Grade 3 or higher, as defined by CTCAE v4.0

SECONDARY OUTCOMES:
Clinical abscopal effect as assessed by number of unradiated lesions with response per RECIST 1.1. | 12 weeks
  Number of lesions that are not targeted by SBRT with any response as defined by RECIST 1.1 criteria. Complete response (CR) = disappearance of all target lesions and normalization of tumor marker levels; Partial response (PR) = decrease from baseline >= 30% in the sum of the longest diameter of all target lesions.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Song, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (2):
- United States (2):
  - Johns Hopkins Bayview, Baltimore, Maryland
  - The Sidney Kimmel Comprehensive Cancer Center at The Johns Hopkins University, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No